CLINICAL TRIAL: NCT05870800
Title: Phase II Open-label Trial of Neoadjuvant Immunotherapy (Atezolizumab) in Combination With CAPOX for Resectable Non-metastatic Proficient Mismatch Repair (pMMR) Colon CancER: NICER Study
Brief Title: Phase II Open-label Trial of Neoadjuvant Immunochemotherapy for Resectable Non-metastatic Colon cancER: NICER
Acronym: NICER
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Atif Iqbal, Associate Professor, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-52907
Record Dates: First submitted 2023-04-11; First posted 2023-05-23 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Stage I Colon Cancer; Stage II Colon Cancer; Stage III Colon Cancer
Keywords: Non-metastatic resectable colon cancer
MeSH Terms: conditions — Colonic Neoplasms | interventions — atezolizumab; Injections; Capecitabine; Oxaliplatin; Leucovorin; Fluorouracil

STUDY DESIGN:
Intervention Model Description: Phase II open-label trial of neoadjuvant CAPOX chemotherapy with Atezolizumab followed by surgery for patients with localized resectable pMMR adenocarcinoma of the colon
Masking Description: Open label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Neoadjuvant Therapy Arm (Experimental): Subjects will receive 4 cycles of neoadjuvant atezolizumab in combination with 4 cycles of CAPOX before standard of care surgical resection. After surgery, patients who are still considered high risk for recurrence (per the treating medical oncologist) will be offered adjuvant therapy.
  Interventions: Drug: Tecentriq 1200 MG in 20 ML Injection + Capecitabine 1000 mg/m2 + Oxaliplatin 130 mg/m2; Drug: Oxaliplatin injection 85mg/m2 + Leucovorin 400mg/m2 + 5-Fluorouracil 2400mg/m2; Drug: Oxaliplatin 130mg/m2 + Capecitabine 1000mg/m2

INTERVENTIONS:
Drug: Tecentriq 1200 MG in 20 ML Injection + Capecitabine 1000 mg/m2 + Oxaliplatin 130 mg/m2 — Enrolled Participant will receive 4 cycles of neoadjuvant Atezolizumab (Tecentriq) followed by CAPOX chemotherapy prior to surgery. Each cycle is every 3 weeks. (12 weeks)
  Other Names: Neoadjuvant Chemoimmunotherapy
Drug: Oxaliplatin injection 85mg/m2 + Leucovorin 400mg/m2 + 5-Fluorouracil 2400mg/m2 — After Surgery, if patients are still considered at high risk (per treating investigator) subjects will be eligible to receive adjuvant chemotherapy with mFOLFOX6 Q2 weeks x 6 cycles (12 weeks) or CAPOX Q3 weeks x 4 cycles (12 weeks)
  Other Names: mFOLFOX6
Drug: Oxaliplatin 130mg/m2 + Capecitabine 1000mg/m2 — After Surgery, if patients are still considered at high risk (per treating investigator) subjects will be eligible to receive adjuvant chemotherapy with mFOLFOX6 Q2 weeks x 6 cycles (12 weeks) or CAPOX Q3 weeks x 4 cycles (12 weeks)
  Other Names: CAPOX

SUMMARY:
This is a Phase II open-label trial of neoadjuvant immunochemotherapy with Atezolizumab and CAPOX followed by surgery and potentially adjuvant chemotherapy for patients with localized resectable pMMR adenocarcinoma of the colon with a target accrual of 28 patients. The investigators will explore if appropriately timed neoadjuvant CAPOX with anti-PD-L1 mAb (Atezolizumab) can be administered safely and feasibly, and that this combination will lead to improved clinical response associated with enhanced numbers of immune cells in surgically resected colon tumors. Patients will receive 4 cycles of atezolizumab in combination with 4 cycles of CAPOX (atezolizumab will be administered prior to chemotherapy) before standard of care surgical resection. Following surgery, patients still considered to be at high-risk of recurrence (per SOC guidelines) will receive further adjuvant chemotherapy (mFOLFOX6 or CAPOX), based on the discretion of the treating oncologist/investigator. Circulating tumor DNA (ctDNA) dynamic change status will be analyzed through collection of blood samples throughout different stages of the patient's neoadjuvant treatment regimen (baseline, pre-neoadjuvant therapy, mid-neoadjuvant, post-neoadjuvant therapy, and during postoperative period) as a marker of early read on efficacy.

The end of the study for each patient enrolled will be at the 6 month postoperative visit.

On Study Protocol: Patients will be followed up for an efficacy follow-up phase during the first 6 months after surgery (week 2 & months 3, 6 visits). All assessments beyond the 6 month visit will be performed under standard of care surveillance office visits.

Off Study Protocol: Thereafter they will enter a survival follow-up phase per standard of care protocols. Patients will be seen every 6 months starting at month 12 until month 36. All collection of research-specific assessments including whole blood, stool collection and quality of life questionnaires will be optional beyond the 6 month postop visit (months 12-36).

DETAILED DESCRIPTION:
This is a Phase II open-label trial of neoadjuvant immunochemotherapy with Atezolizumab + CAPOX chemotherapy followed by surgery and adjuvant chemotherapy (only for high-risk patients) for patients with localized resectable pMMR adenocarcinoma of the colon with a target accrual of 28 patients. The investigational medicinal product (IMP) for this study is atezolizumab. Neoadjuvant CAPOX chemotherapy regimen or category (including rescue medications, premedications), in addition to adjuvant chemotherapy regimens (mFOLFOX6 and CAPOX) are considered non investigational medicinal products (NIMPs).

Please note all RESEARCH ONLY PROCEDURES ARE MARKED WITH A " * " BASELINE VISIT

Once eligibility of potential subjects is confirmed and consent is obtained eligible subjects will undergo the following procedures:

1. Informed Consent *
2. History & Physical exam
3. Vital Signs
4. Assessment of concomitant medications
5. Performance Status (ECOG)
6. PRO/QOL assessments (Research)*
7. Eligibility Assessment*
8. Routine Imaging and Laboratory
9. Blood collection for ctDNA analysis (mandatory) and biobanking (optional)*
10. Stool collection*
11. Urine pregnancy test

NEOADJUVANT THERAPY (RESEARCH) After baseline assessments and eligibility has been confirmed, patients will receive 4 cycles of neoadjuvant immunochemotherapy for a total of 12 weeks. Therapy consists of Atezolizumab in combination with CAPOX (capecitabine + oxaliplatin) before standard-of-care surgical resection. Each cycle of neoadjuvant therapy is 3 weeks. After completion of neoadjuvant therapy, patients will be evaluated during a presurgical evaluation visit for follow-up of any side effects that could potentially arise from therapy and to determine readiness for surgical removal of the tumor (staging evaluation and assessment of response). During this evaluation visit repeat imaging (CT scan or MRI) will be obtained between 2-8 weeks following completion of neoadjuvant therapy. During each cycle the following assessments will be evaluated*:

1. History & Physical exam *
2. Vital Signs *
3. Adverse event assessment*
4. Assessment of concomitant medications *
5. Administration of neoadjuvant therapy with Aztezoluzumab and CAPOX chemotherapy*
6. Routine laboratory assessments*
7. Blood collection for ctDNA analysis (mandatory) and biobanking (optional) during mid-therapy and at conclusion of therapy*
8. Stool collection (after each cycle)*
9. Imaging for disease restaging and therapy response (CT or MRI) of abdomen and pelvis will be obtained after neoadjuvant therapy (2-4 weeks after neoadjuvant therapy)

   * *All assessments for this visit are considered research.

SURGERY Surgical removal of the tumor will be performed per standard-of-care practices. Tumor sample will be obtained per standard of care procedure and will be used after final diagnosis by pathology.

POSTOPERATIVE FOLLOW-UP AND ADJUVANT CHEMOTHERAPY Efficacy Follow-up phase (week 2, month 3 & month 6) Long-term (survival) Follow-up phase (Months 12-36)

Following surgery, patients will enter an efficacy follow-up phase (initial 6 months) and a long-term (survival) follow-up phase (months 12-36). Patients still considered to be at high risk of recurrence (per NCCN guidelines) will receive further adjuvant chemotherapy based on protocol and the discretion of the treating oncologist/investigator.

EFFICACY FOLLOW-UP PHASE ( Week 2 postop and Months 3, 6) Patients will be followed up for an efficacy follow-up phase during first 2 weeks postop and months 3 and 6 and will complete the following assessments:

1. History & Physical exam
2. Vital Signs
3. Adverse event assessment*
4. Assessment of concomitant medications
5. Quality of life assessments (satisfaction survey at week 2 and month 3 only)*
6. Vital status update*
7. Assessment of adjuvant therapy*
8. Blood collection for ctDNA analysis and biobanking* (ctDNA blood draw only at week 2 visit)
9. Stool collection *
10. Adjuvant chemotherapy with standard of care chemotherapy (ONLY FOR HIGH-RISK PATIENTS)
11. Laboratory analysis (CEA,CBC & Chemistry panel)(3 & 6 months only)
12. Standard of care imaging (6 months only)

LONG TERM/ SURVIVAL FOLLOW-UP PHASE Patients will be followed up for an long-term (survival) follow-up phase during months 12, 18, 24, 30, and 36 and will complete the following assessments:

1. History & Physical exam
2. Vital Signs
3. Adverse event assessment*
4. Assessment of concomitant medications
5. Quality of life assessments*
6. Vital status update*
7. Blood collection for biobanking (these samples are optional) *
8. Stool collection *
9. Standard of care imaging

Research procedures:

1. Blood and stool samples will be collected for ctDNA analysis (mandatory) and for banking (optional) at baseline and throughout different stages of the study for future exploratory analysis. The optional blood samples will be stored at Baylor College of Medicine main campus in the ABBR (Alkek Building for Biomedical Research) laboratory and kept for up to 10 years. The purpose of biobanking these samples is for future exploratory research analyses based on future available funding. Stool sample collection kits will be provided to participating subjects which they will be shipping back to our site and collected at several timepoints for storage and future use. In the future stool samples may be used for metabolomic and proteomic profiling. (Costs of shipping back stool kits will be covered by site/sponsor).
2. Quality of life (QOL) outcomes will be obtained through patient- reported outcome (PRO) questionnaires (approx. duration: ~10-20 min per visit) PRO data will be collected through use of the following instruments: MD Anderson Symptom Inventory (MDASI), QLQ C30, and a satisfaction survey. All patients will complete the MDASI, QLQ-C30, and questionnaires at the following timepoints: baseline, after neoadjuvant therapy completion, postoperatively on week 2, months 3, 6, 12, 18, 24, 30, 36. The satisfaction survey will be only collected at week 2 and month 3.
3. Banking procedures: A proper IRB submission will be submitted for request of historic sample controls to previously biobanked specimens within Baylor's biobanks. Historic samples will be deidentified and will be used for comparison. An attempt will be made to match demographics and tumor site but this comparison is going to be used only as an exploratory endpoint.
4. Storage of Data: Each patient will have their own research binder in which research data will be collected. Each subject will be assigned a unique study number ID and will be used throughout the patient's participation. No personal data will be used to identify patients, only the study ID will be used for confidentiality purposes. Data will be captured manually in the patient's binder and electronically in Oncore using study ID number only. Subject binder will be stored in a locked cabinet on the 7th floor at the McNair campus. Only authorized personnel will have access to patient's binder. Information from medical chart that will be used includes: demographic data, concomitant medications, vital signs, medical history, laboratory results, imaging results, notes from office visits, surgery notes, operative notes, progress notes, pathology reports. No information will be shared with any third parties.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form
* Age ≥18 years at time of signing Informed Consent Form
* Ability to comply with the study protocol
* MSS or pMMR tumor determined by local CLIA-certified PCR or IHC testing respectively.
* Histologically or cytologically confirmed resectable non-metastatic adenocarcinoma of the colon.
* The distal extent of the tumor must be ≥12 cm from the anal verge on pre-surgical endoscopy and/or imaging (i.e., excluding rectal adenocarcinomas warranting treatment with chemoradiation). If the patient did not undergo a pre-surgical endoscopy, then the distal extent of the tumor must be ≥12 cm from the anal verge as determined by surgical examination or pre-operative imaging.
* One or more of the following high-risk features:

  * High CEA levels (>5 ng/ml in non-smoker patients , >10ng/ml in smoker patients)
  * Low Lymphocyte-to-monocyte Ratio (<2.38)
  * Poor grade of tumor differentiation
  * Evidence of Lymphovascular Invasion
  * Evidence of Perineural Invasion
  * CT evidence of T3 orT4 disease w/ ≥4 cm tumor longitudinal diameter
  * CT evidence of regional lymphadenopathy
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-1
* Adequate hematologic and end-organ function, defined by the following laboratory test results, obtained within 14 days prior to initiation of study treatment:

  * ANC ≥ 1.5 x 10*9/L (1500/mL) without granulocyte colony-stimulating factor support
  * Lymphocyte count ≥ 0.5 x 10*9/L (500/µL)
  * Platelet count ≥100 x 10*9/L (100,000/µL) without transfusion
  * Hemoglobin ≥ 9 g/L (9 g/dL) Patients may be transfused to meet this criterion.
  * AST, ALT, and alkaline phosphatase (ALP) ≤ 2.5 x upper limit of normal (ULN)
  * Serum bilirubin ≤ 1.5 x ULN with the following exception:

Patients with known Gilbert disease: serum bilirubin ≤ 3 x ULN

* Serum creatinine ≤1.5 x ULN or Creatinine clearance ≥ 50 mL/min (calculated using the Cockcroft-Gault formula)
* Serum albumin ≥ 25 g/L (2.5 g/dL)
* For patients not receiving therapeutic anticoagulation: INR or aPTT ≤ 1.5 x ULN

  * For patients receiving therapeutic anticoagulation: stable anticoagulant regimen
  * Negative hepatitis B surface antigen (HBsAg) test at screening
  * Negative hepatitis C virus (HCV) antibody test at screening, or positive HCV antibody test followed by a negative HCV RNA test at screening The HCV RNA test must be performed for patients who have a positive HCV antibody test.
  * Negative HIV test at screening
  * For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods, and agreement to refrain from donating eggs, as defined below:

Women must remain abstinent or use contraceptive methods with a failure rate of < 1% per year during the treatment period and for 5 months after the final dose of atezolizumab and for 6 months following any of the adjuvant chemotherapy regimens (if applicable) after the final dose of mFOLFOX6 or CAPEOX.Women must refrain from donating eggs during this same period.

A woman is considered to be of childbearing potential if she is postmenarchal, has not reached a postmenopausal state (≥ 12 continuous months of amenorrhea with no identified cause other than menopause), and has not undergone surgical sterilization (removal of ovaries, fallopian tubes and/or uterus) or another cause as determined by the investigator (e.g., Müllerian agenesis). Per this definition, a woman with a tubal ligation is considered to be of childbearing potential. The definition of childbearing potential may be adapted for alignment with local guidelines or requirements.

Examples of contraceptive methods with a failure rate of < 1% per year include bilateral tubal ligation, male sterilization, hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices, and copper intrauterine devices.

The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not adequate methods of contraception. If required per local guidelines or regulations, locally recognized adequate methods of contraception and information about the reliability of abstinence will be described in the local Informed Consent Form.

• For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures, and agreement to refrain from donating sperm, as defined below: With a female partner of childbearing potential who is not pregnant, men who are not surgically sterile must remain abstinent or use a condom plus an additional contraceptive method that together result in a failure rate of <1% per year during the treatment period and for 5 months after the final dose of any chemotherapy regimen. Men must refrain from donating sperm during this same period.

With a pregnant female partner, men must remain abstinent or use a condom during the treatment period and for 5 months after any of the chemotherapy regimens to avoid exposing the embryo.

The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not adequate methods of contraception. If required per local guidelines or regulations, locally recognized adequate methods of contraception and information about the reliability of abstinence will be described in the local Informed Consent Form.

Exclusion Criteria:

* Symptomatic, untreated, or any site actively progressing metastatic disease.
* History of leptomeningeal disease
* Uncontrolled tumor-related pain Patients requiring pain medication must be on a stable regimen at study entry. Presence of any metastatic effusion (pleural, pericardial, ascites)
* Uncontrolled or symptomatic hypercalcemia (ionized calcium > 1.5 mmol/L, calcium > 12 mg/dL or corrected serum calcium > ULN)
* Active or history of autoimmune disease or immune deficiency, including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid antibody syndrome, Wegener granulomatosis, Sjögren syndrome, Guillain-Barré syndrome, or multiple sclerosis (see Appendix 11 for a more comprehensive list of autoimmune diseases and immune deficiencies), with the following exceptions:

Patients with a history of autoimmune-related hypothyroidism who are on thyroid-replacement hormone are eligible for the study.

Patients with controlled Type 1 diabetes mellitus who are on an insulin regimen are eligible for the study.

Patients with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis are excluded) are eligible for the study provided all of following conditions are met:

* Rash must cover < 10% of body surface area
* Disease is well controlled at baseline and requires only low-potency topical corticosteroids
* There has been no occurrence of acute exacerbations of the underlying condition requiring psoralen plus ultraviolet A radiation, methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, or high-potency or oral corticosteroids within the previous 12 months
* History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography (CT) scan History of radiation pneumonitis in the radiation field (fibrosis) is permitted.

  * Active tuberculosis
  * Significant cardiovascular disease (such as New York Heart Association Class II or greater cardiac disease, myocardial infarction, or cerebrovascular accident) within 3 months prior to initiation of study treatment, unstable arrhythmia, or unstable angina
  * Major surgical procedure, other than for diagnosis, within 4 weeks prior to initiation of study treatment, or anticipation of need for a major surgical procedure during the study
  * History of malignancy other than colon adenocarcinoma within 5 years prior to screening, with the exception of malignancies with a negligible risk of metastasis or death (e.g., 5-year OS rate > 90%), such as adequately treated carcinoma in situ of the cervix, non melanoma skin carcinoma, localized prostate cancer, ductal carcinoma in situ, Stage I uterine cancer or colonic polyps
  * Severe infection within 4 weeks prior to initiation of study treatment, including, but not limited to, hospitalization for complications of infection, bacteremia, or severe pneumonia, or any active infection that could impact patient safety
  * Treatment with therapeutic oral or IV antibiotics within 2 weeks prior to initiation of study treatment Patients receiving prophylactic antibiotics (e.g., to prevent a urinary tract infection or chronic obstructive pulmonary disease exacerbation) are eligible for the study.
  * Prior allogeneic stem cell or solid organ transplantation
  * Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that contraindicates the use of an investigational drug, may affect the interpretation of the results, or may render the patient at high risk from treatment complications
  * Treatment with a live, attenuated vaccine within 4 weeks prior to initiation of study treatment, or anticipation of need for such a vaccine during atezolizumab treatment or within 5 months after the final dose of atezolizumab
  * Current treatment with anti-viral therapy for HBV
  * Synchronous primary rectal and/ or colon cancers or history of prior invasive colon malignancy, regardless of disease-free interval.
  * Treatment with investigational therapy within 28 days prior to initiation of study treatment
  * Prior treatment with CD137 agonists or immune checkpoint blockade therapies, including anti-CTLA-4, anti-PD-1, and anti-PD-L1 therapeutic antibodies
  * Treatment with systemic immunostimulatory agents (including, but not limited to, interferon and interleukin 2 [IL-2]) within 4 weeks or 5 half-lives of the drug (whichever is longer) prior to initiation of study treatment
  * Treatment with systemic immunosuppressive medication (including, but not limited to, corticosteroids, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-TNF- agents) within 2 weeks prior to initiation of study treatment, or anticipation of need for systemic immunosuppressive medication during study treatment, with the following exceptions:

Patients who received acute, low-dose systemic immunosuppressant medication or a one-time pulse dose of systemic immunosuppressant medication (e.g., 48 hours of corticosteroids for a contrast allergy) are eligible for the study.

Patients who received mineralocorticoids (e.g., fludrocortisone), corticosteroids for chronic obstructive pulmonary disease (COPD) or asthma, or low-dose corticosteroids for orthostatic hypotension or adrenal insufficiency are eligible for the study.

* History of severe allergic anaphylactic reactions to chimeric or humanized antibodies or fusion proteins
* Known hypersensitivity to Chinese hamster ovary cell products or to any component of the atezolizumab formulation
* Known allergy or hypersensitivity to any component of the CAPOX or mFOLFOX6 chemotherapy formulations
* Pregnancy or breastfeeding, or intention of becoming pregnant during study treatment or within 5 months for Atezolizumab and 6 months for any chemotherapy regimen after the final dose of study treatment Women of childbearing potential must have a negative serum pregnancy test result within 14 days prior to initiation of study treatment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2025-06-15 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Determine the rate of tumor regression grade 1 (<10% viable cancer cells) to neoadjuvant immunotherapy and chemotherapy in resectable (non-metastatic) pMMR colon cancer, assessed in the resection specimen. | 3-5 months
  The primary outcome will be evaluated using the modified Ryan scoring system to score tumor regression grades (TRGs) in the surgical specimen. Scores will be assessed by dedicated study pathologists.
  Success is defined as TRG-0 or TRG-1(<10% viable cancer cells). Efficacy-evaluable participants who do not go to surgery, perhaps due to clinical progression, will be counted as a failure.

SECONDARY OUTCOMES:
Complete pathologic response (TRG-0) to neoadjuvant immunochemotherapy or not. | 36 months
  The investigators will estimate the rate of tumor regression grade (TRG) 0/1 and corresponding exact 95% confidence interval (Wilson method) in the 'efficacy' population. The rate will be compared to the null value of 1% using an exact binomial test with a 5% one-sided significance level. With N=25 efficacy evaluable participants, the investigators will need to see at least 2 grade 0/1 tumor regressions in order to reject the null hypothesis.
R0 resection and number of lymph nodes harvested after neoadjuvant combination CAPOX / Atezolizumab | 3-4 months
  R0 resection rate will be summarized as described for the primary endpoint.
Utilize dynamic changes in ctDNA as an early assessment tool on therapy efficacy. Analysis of ctDNA status to evaluate incidence and changes in surrogate ctDNA biomarker presence. | 36 months
  CtDNA dynamic changes as an early assessment on efficacy. Analysis of ctDNA status (pre-neoadjuvant therapy, mid-neoadjuvant therapy, post- neoadjuvant therapy and postoperative) correlating ctDNA with outcomes and to evaluate incidence and changes in surrogate ctDNA biomarker presence.
Occurrence of any grade 3 or greater adverse events possibly, probably or definitively related to the neoadjuvant CAPOX / Atezolizumab combination | 3-12 months
  This study will utilize the CTCAE (NCI Common Terminology Criteria for Adverse Events) Version 5.0 for toxicity and Serious Adverse Event reporting, with the exception of skin- or nail-related toxicities, which will be graded using CTCAE version 5.0 with modifications. Treatment emergent AE's (grade 3 or greater), will be tabulated with counts of AE's at each grade, as well as counts of participants experiencing any grade 3 or greater treatment emergent AE.
Quality of life as assessed by European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) | 36 months
  QoL scores and patient satisfaction results will be computed using standard guidelines and displayed graphically as spaghetti plots.
  QLQ-C30 scores range from 0 to 100, with higher scores indicating higher/better functioning and higher/better global health status/QoL but lower/worse symptom burden.
Quality of life as assessed by MD Anderson Symptom Inventory (MDASI) | 36 months
  QoL scores and patient satisfaction results will be computed using standard guidelines and displayed graphically as spaghetti plots.
  The M. D. Anderson Symptom Inventory (MDASI) is a brief, patient-reported outcome measure of the impact and severity of 13 cancer-related symptoms that are common across all cancer types. The MDASI score goes from 0 (symptom has not been present) to 10 (the symptom is as worse as it could be) for each item. Higher score means worse outcome.
Delay in surgery after neoadjuvant therapy by more than 12 weeks (84 days) or no | 3-24 months
  Complete surgical resection rates (R0) will be monitored in these patients and if the R0 resection rate is numerically lower than the historical average of ~73% noted in the literature, further analysis of these cases would be performed to ensure that this was not attributed to the delay caused by neoadjuvant therapy.
Rate of treatment acceptance measured by a patient satisfaction questionnaire (PSQ) result at specified time points. | 6-12 months
  An in-house patient satisfaction questionnaire (PSQ) results will be computed using standard guidelines and displayed graphically as spaghetti plots.
  The patient satisfaction questionnaire is a brief, in house, patient satisfaction questionnaire to assess the rate of patient satisfaction, tolerance and acceptance of neoadjuvant treatment used during the study. It includes a brief 10-question assessment and score goes from 0 (not satisfied at all) to 10 (very satisfied).
Overall Survival (OS)- Post-surgery times to event | 36 months
  Post-surgery times to event (OS) will be measured in months throughout the duration of the study (36 months).
  Overall survival (OS) is the time from surgery to death from any cause, regardless of disease recurrence (safety population).
  OS will be summarized by Kaplan-Meier curves, with estimates of median time to event (95% CI by log-log transform), and selected time-specific survival rates (95% CI).
Relapse-free survival (RFS)- Post-surgery times to event | 36 months
  Post-surgery times to event (RFS) will be measured in months throughout the duration of the study (36 months).
  Relapse-free survival (RFS) is defined as the time from surgery to any event, where an "event" is defined first radiographical or pathological evidence of recurrence of disease (excluding second primary cancers) or death from any cause, whichever comes first.
  RFS will be summarized by Kaplan-Meier curves, with estimates of median time to event (95% CI by log-log transform), and selected time-specific survival rates (95% CI).
Time to first recurrence (TTR) -Post-surgery times to event | 36 months
  Post-surgery times to event (TTR) will be measured in months throughout the duration of the study (36 months).
  Time to first recurrence (TTR) is the time from surgery to first radiological or pathological evidence of recurrence, excluding second primary cancers.
  TTR will be summarized by Kaplan-Meier curves, with estimates of median time to event (95% CI by log-log transform), and selected time-specific survival rates (95% CI).

CONTACTS AND LOCATIONS:
Overall Officials: Atif Iqbal, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No